CLINICAL TRIAL: NCT06869421
Title: Knowledge, Attitude and Awareness of Diabetic Patients on Association Between Oral Health and Diabetes Mellitus
Brief Title: Awareness of Patients Having Diabetes Mellitus About Oral Health
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ayat Gamal-AbdelNaser, PI, Cairo University
Other Study IDs: ACU-Med5
Record Dates: First submitted 2025-03-02; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Awareness
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Questionnaire — group of questions about the predictors (age, type of diabetes, level of education) and about the outcomes: knowledge and awareness of the link between diabetes and oral health, and attitude towards maintaining their oral health as diabetics

SUMMARY:
Diabetic patients will be asked to answer a group of questions about the predictors (age, type of diabetes, level of education) and about the outcomes [knowledge and awareness of the link between diabetes and oral health, and attitude towards maintaining their oral health as diabetics.

DETAILED DESCRIPTION:
The study will recruit patients having diabetes mellitus; where they will be asked to answer a questionnaire after obtaining an informed consent. Diabetic patients will be asked to answer a group of questions about the predictors (age, type of diabetes, level of education) and about the outcomes knowledge and awareness of the link between diabetes and oral health, and attitude towards maintaining their oral health as diabetics.

ELIGIBILITY:
Inclusion Criteria:

* aged at least 18 years and being diagnosed with diabetes mellitus

Exclusion Criteria:

* individuals who refuse to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients having diabetes mellitus
Sampling Method: Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
knowledge and awareness of the link between diabetes and oral health | 2 months
  questions 1,2,3,5,6,7,9 in questionnaire of knowledge: Diabetes may increase risk of developing oral health problems Diabetes may increase risk of periodontal problems (gum bleeding, teeth mobility, etc) Diabetes may cause reduction in salivary flow Controlling diabetes is important to minimize oral health complications Saliva is important to maintain oral health resistance to disease such as caries and gum inflammation Regular dental visit is more important for diabetic patients than non-diabetics When visiting the dentist, it is important to inform him about my general health including diabetes